CLINICAL TRIAL: NCT05624593
Title: P200TE Agreement and Precision Study
Brief Title: P200TE and Predicate Agreement and Precision Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1088
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Normal; Retina Disease; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Optical Coherence Tomography (OCT) (Other)
  Interventions: Device: P200TE; Device: Predicate

INTERVENTIONS:
Device: P200TE — The P200TE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
Device: Predicate — The predicate device is an optical coherence tomography system intended for in vivo imaging, axial cross-sectional, three-dimensional imaging and measurement of anterior and posterior ocular structures.

SUMMARY:
This study is a prospective comparative, randomized, single center study to assess agreement and precision of the P200TE in comparison to the predicate device in normal subjects, subjects with glaucoma, and subjects with retinal disease.

ELIGIBILITY:
Inclusion Criteria for Normal Group

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects with normal eye examinations in both eyes on the date of the study visit as observed with a 90 diopter lens
4. BCVA 20/40 or better (each eye) on the date of the study visit

Exclusion Criteria for Normal Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
4. Presence of any ocular pathology except for cataract in either eye

Inclusion Criteria for Glaucoma Group

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. BCVA 20/40 or better in the study eye
4. History of Visual field defects within the previous year from the study visit or measured the day of the study visit consistent with glaucomatous optic nerve damage with at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."
5. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   1. Diffuse thinning, focal narrowing, or notching of the neuroretinal rim, especially at the inferior or superior poles with or without disc hemorrhage;
   2. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue

Exclusion Criteria for Glaucoma Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
4. No reliable Humphrey Field Analyzer (HFA) visual field (24-2 Sita Standard or Fast, white on white) result within the past year of the study visit, defined as fixation losses > 33% or false positives > 33%, or false negatives > 33% in the study eye
5. Presence of any ocular pathology except glaucoma in the study eye

Inclusion Criteria for Retina Disease Group

1. Subjects 22 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with retinal disease
4. BCVA 20/400 or better in the study eye
5. Diagnosis of some type of retinal pathology by investigator, may include, but not limited to: Macular Degeneration (including patients with drusen and geographic atrophy and choroidal neovascularization), Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Central Serous Retinopathy and others

Exclusion Criteria for Retinal Disease Group

1. Subjects unable to tolerate ophthalmic imaging
2. Subjects not able to obtain acceptable OCT images due to ocular media opacity or other reasons
3. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
4. Presence of glaucoma or any ocular pathology other than a retinal pathology (e.g., cornea pathology) in the study eye as determined by self report and/or investigator assessment at the study visit;

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Limit of Agreement (LOA) between the P200TE and predicate device measurements of full retinal thickness. | 1 year
Limit of Agreement (LOA) between the P200TE and predicate device measurements of retinal nerve fiber layer thickness (μm). | 1 year
Limit of Agreement (LOA) between the P200TE and predicate device measurements of ganglion cell complex thickness (μm). | 1 year
Limit of Agreement (LOA) between the P200TE and predicate device measurements of optic disc (disc area, rim area, cup-to-disc area, cup-to-disc vertical, cup-to-disc horizontal) | 1 year
Precision between the P200TE and predicate device measurements of full retinal thickness | 1 year
Precision between the P200TE and predicate device measurements of retinal nerve fiber layer thickness. | 1 year
Precision between the P200TE and predicate device measurements of ganglion cell complex thickness | 1 year
Precision between the P200TE and predicate device measurements of optic disc (disc area, rim area, cup-to-disc area, cup-to-disc vertical, cup-to-disc horizontal) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois College of Optometry, Chicago, Illinois, United States